CLINICAL TRIAL: NCT02886169
Title: Effect of Supplementation of a High-fat Meal With Sacha Inchi Oil on Postprandial Metabolic and Inflammatory Responses in Adults With Low Physical Activity and Without Abdominal Obesity
Brief Title: Effectiveness of Sacha Inchi Supplementation on Postprandial Inflammation
Acronym: ESISOPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Icesi (Other)
Collaborators: Universidad de San Buenaventura (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CA051356
Record Dates: First submitted 2016-08-11; First posted 2016-09-01 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Diseases
Keywords: Sacha Inchi; High-fat meal; Postprandial inflammatory responses
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High fat meal with Sacha Inchi (Experimental): Participants will receive 100 g of bread with 70 g of butter (high saturated fat meal) added with 15ml of Sacha Inchi oil and 125ml of coffee with 10g of sugar
  Interventions: Other: High fat meal with Sacha Inchi
- unsupplemented group (Placebo Comparator): Participants will receive 100 g of bread with 70 g of butter (high saturated fat meal) and 125ml of coffee with 10g of sugar
  Interventions: Other: high saturated fat meal

INTERVENTIONS:
Other: High fat meal with Sacha Inchi — Participants will receive 100 g of bread with 70 g of butter (high saturated fat meal) added with 15ml of Sacha Inchi oil and 125ml of coffee with 10g of sugar
  Arms: High fat meal with Sacha Inchi
Other: high saturated fat meal — Participants will receive 100 g of bread with 70 g of butter (high saturated fat meal) and 125ml of coffee with 10g of sugar
  Arms: unsupplemented group

SUMMARY:
The postprandial state increases triglyceride-rich lipoproteins and lipopolysaccharide (LPS) levels, promoting cellular lipids accumulation, insulin resistance, increased inflammatory markers and the formation of foam cells, a situation that can have different effects depending the type of dietary fat and presence of metabolic conditions such as abdominal obesity and insulin resistance.

Given that the diet of the Colombian population is rich in saturated fats, and taking into consideration the general resistance to complex dietary changes, the purpose of this study is to evaluate whether Sacha Inchi oil supplementation of a high-fat meal is effective in reducing levels of biochemical markers of cardiovascular risk in adults with and without abdominal obesity.

DETAILED DESCRIPTION:
Study population:

The sample will be taken from the population of administrative staff and professors of San Buenaventura University of Cartagena. They will be invited to participate adult men aged between 27 and 59 years with and without abdominal obesity.

Sample size:

To calculate the sample size, a statistical formula was used which allows the comparison of two paired means (repeated measures) in 2 groups. Since there may be a substantial degree of correlation between the magnitude of the baseline measurement and the subsequent, It is necessary to correct the formula for the correlation coefficient, that it was estimated, like the standard deviation (SD), from previous experiences.

The minimum number of subjects (n) for each study group was defined according to the estimate for similar studies in design and study variables, considering as main study variable the levels of triglycerides. Considering the following values: Za = 1,64; Z = 1,28; Mde - Mdc = expected minimum difference = 48; Standard deviation of the primary endpoint = 78,6 and a correlation coefficient of 0,6. With these values the n in both groups was 18 subjects. 21 participants with abdominal obesity and 21 without abdominal obesity will be included providing a 20% of losses.

Method:

1. Catchment: The initial selection of potential participants in the study will be made from the review of the lists of administrators and professors at the University of San Buenaventura in Cartagena. From this list will be selected randomly using random numbers of Excel program a total of 100 participants. People who meet the inclusion criteria will be informed of the study and invited to participate by reading and signing informed consent. They will conduct a survey and anthropometric measurements were taken (weight, height, waist circumference).
2. Intervention: Participants will be cited on two occasions, one week apart, in the morning and after fasting for 12 hours, for breakfast and perform blood sampling. Before the intervention the order in which they will receive breakfast (AB or BA) will be drawn. On each occasion three blood samples were taken per participant (fasting, 1 and 4 hours postprandial).
3. Follow up: During the week between the two interventions, participants follow the recommendations to maintain their usual diet.
4. Sampling: The samples will be taken by a clinical laboratory assistant in EDTA tubes and dry tubes. At the laboratory, plasma and serum will be separated by centrifugation. The samples will be stored at -20 ° C until quantification of the variables of interest.
5. Quantification of biochemical variables: lipopolysaccharide (LPS) will be quantified in plasma by the Limulus amebocyte lysate test. The concentrations of glucose, total cholesterol and triglycerides will be quantified by spectrophotometric enzyme assays. Insulin will be measured by immunoassay.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 27 and 59 years.
* Give voluntary, signed informed consent.
* Group A: Be non-obese as defined as Waist circumference < 92 cm (Gallo, 2003)
* Group B: Be obese as defined as Waist circumference > 92 cm
* Physical inactivity (Adults aged 18-64 who do less than 150 minutes of moderate
* intensity aerobic physical activity throughout the week or less than 75 minutes of
* vigorous-intensity aerobic physical activity throughout the week or an equivalent
* combination of moderate- and vigorous-intensity activity).

Exclusion Criteria:

* Individuals with known gastrointestinal, renal or cardiovascular diseases, diabetes mellitus, fat intolerance, or those taking medications known to affect lipid metabolism or fat absorption.

Ages: 27 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Effect of the different meal combinations on change from baseline plasma triglycerides (in mg/dL) at 1 and 4 hours after breakfast | 0, 1 and 4 hours after breakfast

SECONDARY OUTCOMES:
Effect of the different meal combinations on change from baseline plasma Cholesterol (in mg/dL) at 1 and 4 hours after breakfast | 0, 1 and 4 hours after breakfast
Effect of the different meal combinations on change from baseline plasma High density lipoprotein cholesterol (HDL-Cholesterol , in mg/dL) at 1 and 4 hours after breakfast | 0, 1 and 4 hours after breakfast
Effect of the different meal combinations on change from baseline plasma Glucose (in mg/dL) at 1 and 4 hours | 0, 1 and 4 hours after breakfast
Effect of the different meal combinations on change from baseline plasma insulin (in uIU/mL) at 1 and 4 hours | 0, 1 and 4 hours after breakfast
Effect of the different meal combinations on change from baseline plasma Homeostatic model assessment (HOMA index) (in uIU/mL) at 1 and 4 hours | 0, 1 and 4 hours after breakfast
Effect of the different meal combinations on change from baseline plasma Lipopolysaccharides (EU/mL) at 1 and 4 hours | 0, 1 and 4 hours after breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Echeverri, Doctor, Principal Investigator — Icesi University
Locations (1):
- University of San Buenaventura, Cartagena, Departamento de Bolívar, Colombia

IPD SHARING:
Plan to Share IPD: Yes